CLINICAL TRIAL: NCT01721421
Title: Feasibility and Physiological and Nutritional Effects of Extended Treatment Duration in Patients With End-stage Renal Disease on Haemodialysis
Brief Title: Effects of Extended Haemodialysis Treatment Duration in Patients With End-stage Renal Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 11-LL-0505
Record Dates: First submitted 2012-11-01; First posted 2012-11-05 (Estimated); Last update posted 2012-11-05 (Estimated); Status verified 2012-11

CONDITIONS: End Stage Renal Disease
Keywords: haemodialysis; Crossover; Treatment time; nutritional status
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extended Treatment time (Experimental): Extended treatment time of 6 hours
  Interventions: Other: extended treatment time; Other: Standard treatment time
- standard treatment time (Active Comparator): Standard Treatment time of 4 hours
  Interventions: Other: extended treatment time; Other: Standard treatment time

INTERVENTIONS:
Other: extended treatment time — patients receive extended dialysis treatment time time of 6 hours
Other: Standard treatment time

SUMMARY:
Design: Prospective randomised cross-over study. Fifty-two eligible patients will be randomised to a treatment time of either 6 hours or 4 hours for a period of 24 weeks and following a washout period of 4 weeks, switch to the alternative treatment time for an additional 24 weeks.

Aims: To examine the feasibility and effect of extended dialysis treatment time, 6 hours thrice weekly, versus the standard, 4 hours thrice weekly, comparing the differences from baseline in outcome measures over a total 12-month period.

Primary outcome measure

1]Serum albumin

Secondary outcome measures Nutritional status

1. Malnutrition-inflammation score
2. Dietary intake
3. Hand-Grip strength
4. Energy expenditure

Quality of life

1. Patient reported quality of life and
2. time to recovery from dialysis

Serum biomarkers

1. BNP
2. Troponin
3. MCP-1

Others 24- hour Ambulatory blood pressure 24-hour accelerometer

Population: Local haemodialysis population of 1200 patients Eligibility: Minimum 90days on haemodialysis treatment Duration: Fifty-six weeks

ELIGIBILITY:
Inclusion Criteria:

* Dialysis dependant for over 90 days

Exclusion Criteria:

1. Haemodialysis for less than 90 days
2. Patients with anticipated life expectancy less than 6 months secondary to significant morbidity e.g. metastatic malignancy, advanced human immunodeficiency virus
3. Patients with acute liver disease; History of underlying haematological condition;
4. Elective planned change of renal replacement modality within the 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2011-09; Primary Completion 2014-03 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Serum albumin | baseline to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Choi, MBcHB PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom